CLINICAL TRIAL: NCT02047097
Title: A Multicenter, Global, Observational Study to Collect Information on Safety and to Document the Drug Utilization of Tecfidera™ (Dimethyl Fumarate) When Used in Routine Medical Practice in the Treatment of Multiple Sclerosis (ESTEEM)
Brief Title: Dimethyl Fumarate (DMF) Observational Study
Acronym: ESTEEM
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS401
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dimethyl fumarate (DMF): Patients with multiple sclerosis receiving dimethyl fumarate (DMF) under routine clinical care
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — Provided under routine clinical care
  Other Names: Tecfidera; DMF; BG00012

SUMMARY:
The primary objective of the study is to determine the incidence, type, and pattern of serious adverse events (SAEs), including but not limited to infections (including opportunistic infections), hepatic events, malignancies, and renal events, and of adverse events (AEs) leading to treatment discontinuation in patients with MS treated with dimethyl fumarate (DMF). Secondary objectives of this study in this population are as follows: To determine dimethyl fumarate (DMF) prescription and utilization patterns in routine clinical practice in patients with multiple sclerosis (MS); To assess the effectiveness of dimethyl fumarate (DMF) on multiple sclerosis (MS) disease activity and disability progression in routine clinical practice as determined by the Expanded Disability Status Scale (EDSS) score and multiple sclerosis (MS) relapse information; and To assess the effect of dimethyl fumarate (DMF) on health-related quality of life, healthcare resource consumption, and work productivity.

DETAILED DESCRIPTION:
Patients aged 12 to under 18 may be included where enrollment of pediatric patients in this study is considered observational and is permissible by local regulations.

ELIGIBILITY:
Key Inclusion Criteria:

- Patients with multiple sclerosis (MS) who are newly initiating treatment with dimethyl fumarate (DMF) under routine clinical care are eligible to participate in the study.

Key Exclusion Criteria:

* Patients with previous exposure to dimethyl fumarate (DMF), Fumaderm (fumaric acid esters), or compounded fumarates.
* Patients participating in other clinical studies.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine clinical care for Multiple Sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 5487 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The number of participants that experience Adverse Events (AEs) that lead to discontinuation of dimethyl fumarate (DMF) | Up to 5 years
The number of participants that experience Serious Adverse Events (SAEs) | Up to 5 years

SECONDARY OUTCOMES:
Duration of dimethyl fumarate (DMF) use | Up to 5 years
dimethyl fumarate (DMF) dosing frequency | Up to 5 years
Primary reasons for discontinuation of dimethyl fumarate (DMF) use | Up to 5 years
Frequency of relapses over time | Up to 5 years
Disease progression as measured by Expanded Disability Status Scale (EDSS) over time | Up to 5 years
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist. Participants with confirmed progression of disability in EDSS physical functional system scores will be defined as those who meet one of the following criteria: an increase of ≥ 1 point from baseline system score of ≥ 1 or an increase of ≥ 2 points from baseline system score of 0 in at least 2 physical functional systems, or an increase of ≥ 2 points from baseline system score of ≥ 1 or an increase of ≥ 3 points from baseline system score of 0 in any 1 physical functional system. Worsening must be confirmed on a subsequent examination using the same criterion in the same functional system(s) at least 6 months later.
Multiple Sclerosis Impact Scale-29 Items (MSIS-29) physical multiple sclerosis (MS) impact score | Up to 5 years
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a patient-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a patient's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.
Multiple Sclerosis Impact Scale-29 Items (MSIS-29) psychological multiple sclerosis (MS) impact score | Up to 5 years
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a patient-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a patient's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.
EuroQol-5 Dimensions (5 Level) (EQ-5D-5L) index score | Up to 5 years
  Descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension.
EuroQol Visual Analogue Scale (EQ VAS) (0-100 scale) | Up to 5 years
  Standard vertical 20 cm visual analogue scale (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state (often referred to as page 3 of the EQ-5D questionnaire)
Modified Fatigue Impact Scale-5 (MFIS-5) total score | Up to 5 years
  MFIS-5 is a modified form of the Fatigue Impact Scale that consists of five questions that assess the impact of fatigue on physical, cognitive, and psychosocial functioning, with five response levels ranging from 0 ("Never") to 4 ("Almost always"). Total scores range from 0 to 20, with higher scores representing a greater impact of fatigue.
Work Productivity and Activity Impairment questionnaire: Multiple Sclerosis, Version 2.0 (WPAI-MS) impairment percentages | Up to 5 years
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Health Care Resource Consumption Questionnaire | Up to 5 years
  The Health Care Resource Consumption questionnaire is a survey that asks patients how MS affects their use of healthcare services and the impact it has on particular areas of their life (including number of hospitalizations [MS-related, non-MS related, relapse-related, resulting in steroid use], MS-related emergency room visits, MS-related neurologist visits, visits to other health care professionals for MS-related and other reasons).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (412):
- United States (146):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Sites, Fullerton, California
  - Research Site, Hanford, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, San Francisco, California
  - Research Site, Santa Ana, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Derby, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Norwich, Connecticut
  - Research Site, Dover, Delaware
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Sites, Boca Raton, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Sites, Lighthouse PT, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Sites, Atlanta, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Herrin, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Elkhart, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Henderson, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Hammond, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Rockport, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Glen Burnie, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Foxborough, Massachusetts
  - Research Site, Jamaica Plain, Massachusetts
  - Research Site, Lexington, Massachusetts
  - Research Site, Wellesley, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, West Bloomfield, Michigan
  - Research Site, Edina, Minnesota
  - Research Sites, Minneapolis, Minnesota
  - Research Site, Ocean Springs, Mississippi
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Great Falls, Montana
  - Research Sites, Lincoln, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Wahoo, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Concord, New Hampshire
  - Research Site, Audubon, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, Livingston, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Stratford, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, West Long Branch, New Jersey
  - Research Site, Albany, New York
  - Research Site, Cedarhurst, New York
  - Research Site, East Meadow, New York
  - Research Site, Kingston, New York
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, Plainview, New York
  - Research Site, Syracuse, New York
  - Research Site, Asheville, North Carolina
  - Research Sites, Charlotte, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Sites, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Centerville, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Allentown, Pennsylvania
  - Research Site, Greensburg, Pennsylvania
  - Research Site, Meadowbrook, Pennsylvania
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Natrona Heights, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Colleyville, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Green Bay, Wisconsin
  - Research Site, La Crosse, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Neenah, Wisconsin
  - Research Site, Waukesha, Wisconsin
- Argentina (12):
  - Research Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Vicente López, Buenos Aires
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Salta
  - Research Site, San Juan
  - Research Site, Santiago del Estero
  - Research Site, Villa Nueva
- Australia (20):
  - Research Site, Camperdown, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Gold Coast, Queensland
  - Research Site, Bedford Park, South Australia
  - Research Site, Kent Town, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Clayton, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Nedlands, Western Australia
- Austria (3):
  - Research Site, Amstetten
  - Research Site, Salzburg
  - Research Site, Vienna
- Canada (15):
  - Research Site, Calgary, Alberta
  - Research Site, Burnaby, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Cambridge, Ontario
  - Research Site, London, Ontario
  - Research Site, Milton, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Gatineau, Quebec
  - Research Sites, Montreal, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Regina, Saskatchewan
- Czechia (7):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Olomouc
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Teplice
- Denmark (5):
  - Research Site, Aarhus C
  - Research Site, Esbjerg
  - Research Site, Glostrup Municipality
  - Research Site, Odense C
  - Research Site, Sønderborg
- France (13):
  - Research Site, Montluçon, Allier
  - Research Site, Mulhouse, Haut Rhin
  - Research Site, Toulouse, Haute Garonne
  - Research Site, Pringy, Haute Savoie
  - Research Site, Rueil-Malmaison, Hauts De Seine
  - Research Site, Dax, Landes
  - Research Site, Agen, Lot Et Garonne
  - Research Site, Perpignan, Pyrenees Orientales
  - Research Site, Bron, Rhone
  - Research Site, La Roche-sur-Yon, Vendee
  - Research Site, Épinal, Vosges
  - Research Site, Gonesse
  - Research Site, Rambouillet
- Germany (68):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Heidenheim, Baden-Wurttemberg
  - Research Site, Ladenburg, Baden-Wurttemberg
  - Research Site, Mannheim, Baden-Wurttemberg
  - Research Site, Ravensburg, Baden-Wurttemberg
  - Research Site, Singen, Baden-Wurttemberg
  - Research Site, Sinsheim, Baden-Wurttemberg
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, Ulm, Baden-Wurttemberg
  - Research Site, Alzenau in Unterfranken, Bavaria
  - Research Site, Bayreuth, Bavaria
  - Research Site, Bogen, Bavaria
  - Research Site, Erlangen, Bavaria
  - Research Site, Landshut, Bavaria
  - Research Site, Munich, Bavaria
  - Research Site, Neuburg am Inn, Bavaria
  - Research Site, Nuremberg, Bavaria
  - Research Site, Regensburg, Bavaria
  - Research Site, Unterhaching, Bavaria
  - Research Site, Wolfratshausen, Bavaria
  - Research Site, Würzburg, Bavaria
  - Research Site, Butzbach, Hesse
  - Research Site, Eltville, Hesse
  - Research Site, Erbach im Odenwald, Hesse
  - Research Site, Eschwege, Hesse
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Gelnhausen, Hesse
  - Research Site, Giessen, Hesse
  - Research Site, Gladenbach, Hesse
  - Research Site, Kassel, Hesse
  - Research Site, Wiesbaden, Hesse
  - Research Site, Buchholz, Lower Saxony
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Oldenburg, Lower Saxony
  - Research Site, Stade, Lower Saxony
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Bad Honnef, North Rhine-Westphalia
  - Research Site, Bergisch Gladbach, North Rhine-Westphalia
  - Research Site, Bielefeld, North Rhine-Westphalia
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Bonn, North Rhine-Westphalia
  - Research Site, Cologne, North Rhine-Westphalia
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Hagen, North Rhine-Westphalia
  - Research Site, Remscheid, North Rhine-Westphalia
  - Research Site, Siegen, North Rhine-Westphalia
  - Research Site, Willich, North Rhine-Westphalia
  - Research Site, Wuppertal, North Rhine-Westphalia
  - Research Site, Frankenthal, Rhineland-Palatinate
  - Research Site, Kandel, Rhineland-Palatinate
  - Research Site, Katzenelnbogen, Rhineland-Palatinate
  - Research Site, Rülzheim, Rhineland-Palatinate
  - Research Site, Trier, Rhineland-Palatinate
  - Research Site, Chemnitz, Saxony
  - Research Site, Görlitz, Saxony
  - Research Site, Leipzig, Saxony
  - Research Site, Wermsdorf, Saxony
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Eisenach, Thuringia
  - Research Site, Erfurt, Thuringia
  - Research Site, Jena, Thuringia
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Neusäß
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Eger
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Szeged
  - Research Site, Tatabánya
  - Research Site, Zalaegerszeg
- Research Site, Dublin, Ireland
- Italy (24):
  - Research Site, Torrette, Ancona
  - Research Site, Montichiari, Brescia
  - Research Site, Pozzilli, Isernia
  - Research Site, Legnano, Milano
  - Research Site, Fidenza, Parma
  - Research Site, Orbassano, Torino
  - Research Site, Gallarate, Varese
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Cagliari
  - Research Site, Catanzaro
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pordenone
  - Research Site, Reggio Emilia
  - Research Site, Roma
- Netherlands (13):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Geldrop
  - Research Site, Geleen
  - Research Site, Hoorn
  - Research Site, Leeuwarden
  - Research Site, Leiden
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Tilburg
  - Research Site, Venlo
- New Zealand (3):
  - Research Site, Christchurch
  - Research Site, Dunedin
  - Research Site, Hamilton
- Norway (2):
  - Research Site, Bodø
  - Research Site, Namsos
- Poland (17):
  - Research Site, Ochojec, Katowice
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gmina Końskie
  - Research Site, Grudziądz
  - Research site, Głogów Małopolski
  - Research site, Katowice
  - Research Site, Katowice
  - Research site, Konstancin-Jeziorna
  - Research Site, Krakow
  - Research site, Krakow
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Zabrze
- Portugal (8):
  - Research Site, Amadora
  - Research Site, Braga
  - Research Site, Guimarães
  - Research Site, Matosinhos Municipality
  - Research Site, Penafiel
  - Research Site, Santarém
  - Research Site, Viana do Castelo
  - Research Site, Vila Nova de Gaia
- Puerto Rico (2):
  - Research Site, Guaynabo
  - Research Site, San Juan
- Slovakia (8):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research site, Martin
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Ružomberok
  - Research Site, Trenčín
  - Research Site, Trnava
- Spain (16):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Badalona, Barcelona
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Santander, Cantabria
  - Research Site, Santiago de Compostela, La Coruña
  - Research Site, Gijón, Principality of Asturias
  - Research Site, Santa Cruz de Tenerife, Tenerife
  - Research Site, Alzira, Valencia
  - Research Site, Ávila
  - Research Site, Cadiz
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Murcia
  - Research Site, Pontevedra
- Switzerland (3):
  - Research Site, Bern
  - Research Site, Lausanne
  - Research Site, Lugano
- United Kingdom (19):
  - Research Site, Bristol, Avon
  - Research Site, Exeter, Devon
  - Research Site, Plymouth, Devon
  - Research Site, Torquay, Devon
  - Research Site, Salford, Greater Manchester
  - Research Site, Basingstoke, Hampshire
  - Research Site, Southampton, Hampshire
  - Research Site, Leicester, Leicestershire
  - Research Site, Edinburgh, Lothian Region
  - Research Site, Liverpool, Merseyside
  - Research Site, Norwich, Norfolk
  - Research Site, Nottingham, Nottinghamshire
  - Research Site, Glasgow, Strathclyde
  - Research Site, Dundee, Tayside Region
  - Research Site, Newcastle upon Tyne, Tyne & Wear
  - Research Site, Birmingham, West Midlands
  - Research Site, Leeds, West Yorkshire
  - Research Site, Belfast
  - Research Site, Swansea

REFERENCES:
- [Derived] Pandey KS, Giles K, Balashov K, Macdonell R, Windsheimer J, Martinez M, Bozin I, Raynaud S, Scaramozza M, Mokliatchouk O, Sun Z, Belviso N, Sato Y, Lin X, Okai A. Long-Term Safety and Effectiveness of Dimethyl Fumarate in Patients with Multiple Sclerosis Treated in Routine Medical Practice: Final Analysis of the ESTEEM Study. Neurol Ther. 2025 Feb;14(1):243-260. doi: 10.1007/s40120-024-00680-z. Epub 2024 Dec 14. PMID 39673658
- [Derived] Mao-Draayer Y, Bar-Or A, Balashov K, Foley J, Smoot K, Longbrake EE, Robertson D, Mendoza JP, Lewin JB, Everage N, Bozin I, Lyons J, Mokliatchouk O, Bame E, Giuliani F. Real-World Safety and Effectiveness of Dimethyl Fumarate in Patients with MS: Results from the ESTEEM Phase 4 and PROCLAIM Phase 3 Studies with a Focus on Older Patients. Adv Ther. 2025 Jan;42(1):395-412. doi: 10.1007/s12325-024-03047-w. Epub 2024 Nov 21. PMID 39570545
- [Derived] Williams MJ, Amezcua L, Chinea A, Cohan S, Okai A, Okuda DT, Vargas W, Belviso N, Bozin I, Jiang X, Lewin JB, Lyons J, Shen C, England SM, Grimes N. Real-World Safety and Effectiveness After 5 Years of Dimethyl Fumarate Treatment in Black and Hispanic Patients with Multiple Sclerosis in ESTEEM. Neurol Ther. 2023 Oct;12(5):1669-1682. doi: 10.1007/s40120-023-00517-1. Epub 2023 Jun 24. PMID 37354276